CLINICAL TRIAL: NCT07375875
Title: Strategies to Minimize the Risk for Insulin Induced Hypertrophy and Its Related Consequences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Marwa Fathallah Mostafa, professor of critical and emergency nursing, Mansoura University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 0307290 Faculty of medicine, A
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Insulin Dependent Diabetes Mellitus
Keywords: Strategies; Insulin; Injection; Hypertrophy; Map
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance; Hypertrophy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group(1) (Active Comparator): Insulin site injection map
  Interventions: Procedure: Group(1) Insulin site injection map
- Group two (No Intervention): Routine hospital care with continuous follow up

INTERVENTIONS:
Procedure: Group(1) Insulin site injection map — The intervention group participants attended a structured educational session focused on strategies to reduce the risk of insulin-induced hypertrophy and its associated consequences, either individually or in small groups . The session included: appropriate insulin injection techniques, since repeated trauma is the main cause of hypertrophy, the researchers explained "standardized rotation protocols and insulin injection sites map"
  Arms: Group(1)

SUMMARY:
Hypertrophy caused by insulin has effects that extend beyond just aesthetic concerns. Innovative methods have shown potential in decreasing the chances of hypertrophy and its related issues, including the development of detailed diagrams of insulin injection locations and tailored rotation plans. This study aimed to assess the impact of a novel insulin injection sites map (digital or physical) on the incidence of insulin-induced hypertrophy, adherence to rotation protocols, glycemic control, and patient experience among diabetes patients treated with insulin between study and control group along six months of follow up

DETAILED DESCRIPTION:
Patients on long-term insulin therapy frequently experience significant side effect of insulin-induced hypertrophy, particularly lipohypertrophy (LH).Nurses play a crucial role as direct care providers and educators for diabetes patients, ensuring the safe administration of insulin and preventing insulin-related hypertrophy. This research aims to explore and evaluate innovative mapping methods for insulin injection locations due to the rising prevalence of diabetes in Egypt and the United States, alongside the considerable effect that insulin-induced hypertrophy has on patient results and healthcare systems

ELIGIBILITY:
Inclusion Criteria:

* • Type 1 or type 2 diabetes mellitus in adults (≥18 years old).

  * Insulin therapy has been administered for a minimum of six months.
  * Self-injecting insulin and assisted injection on a regular basis

Exclusion Criteria:

* Patients with mental illnesses or severe cognitive impairment.

  * Individuals with skin disorders at injection locations such as severe eczema, psoriasis, or infection that could interfere with the evaluation of lipohypertrophy.
  * Women who are lactating or pregnant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Decrease Lipohypertrophy | 6 months
  insulin induced lipohypertrophy

CONTACTS AND LOCATIONS:
Overall Officials: Hala Mohamed Abdelhamed, Assis.prof, Study Director — Faculty of Nursing, Mansoura university; Hoda Eldeeb, Assis.prof, Study Director — Faculty of nursing, ِAlexandria University
Locations (1):
- faculty of nursing, Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] • American Diabetes Association Professional Practice Committee; 6. Glycemic Goals and Hypoglycemia: Standards of Care in Diabetes-2024. Diabetes Care 1 January 2024; 47 (Supplement_1): S111-S125. https://doi.org/10.2337/dc24-S006 • Bavuma, C. M., Musafiri, S., Rutayisire, P. C., Ng'ang'a, L. M., McQuillan, R., & Wild, S. H. (2020). Socio-demographic and clinical characteristics of diabetes mellitus in rural Rwanda: time to contextualize the interventions? A cross-sectional study. BMC endocrine disorders, 20(1), 180. https://doi.org/10.1186/s12902-020-00660-y • Blanchard, J., Ahmed, S., Clark, B., Sanchez Cotto, L., Rangasamy, S., & Thompson, B. (2024). Design and Testing of a Smartphone Application for Real-Time Tracking of CSII and CGM Site Rotation Compliance in Patients With Type 1 Diabetes. Journal of Diabetes Science and Technology, 18(4), 937-945.